CLINICAL TRIAL: NCT00006163
Title: Computer-assisted Diabetes Self-management Interventions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Factorial
Other Study IDs: glasgowr (completed); 35524
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; self-management; randomized trial; RE-AIM evaluation; participation; maintenance; community resources; dietary change
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Community Resources

INTERVENTIONS:
Behavioral: Personalized Self-management
Behavioral: Community Resources

SUMMARY:
This project evaluates the effectiveness of different aspects of a program to assist type 2 diabetes patients with dietary changes. It evaluates the effectiveness of Personalized Self-Management Training and Community Resources support, using a randomized design. This study will also evaluate what percent of patients are willing to participate in such a program, and what percent of primary care physicians are willing to recommend it to their patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Diagnosed for at least one year
* Patient of a primary care provider

Exclusion Criteria:

* No telephone
* Not speaking English

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-09; Study Completion 1999-06

CONTACTS AND LOCATIONS:
Locations (1):
- AMC Cancer Research center, Denver, Colorado, United States

REFERENCES:
- [Background] Glasgow RE, La Chance PA, Toobert DJ, Brown J, Hampson SE, Riddle MC. Long-term effects and costs of brief behavioural dietary intervention for patients with diabetes delivered from the medical office. Patient Educ Couns. 1997 Nov;32(3):175-84. doi: 10.1016/s0738-3991(97)00039-6. PMID 9423499